CLINICAL TRIAL: NCT00739791
Title: Pilot Trial of Gene Expression Modulation by Intervention With Nutrition and Lifestyle
Brief Title: Nutrition and Lifestyle Changes in Patients With Previously Untreated Stage I or Stage II Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Peter R. Carroll, UCSF Helen Diller Family Comprehensive Cancer Center
Purpose: Treatment
Other Study IDs: CDR0000612335; UCSF-H5664-25348; UCSF CC#04553
Record Dates: First submitted 2008-08-21; First posted 2008-08-22 (Estimated); Last update posted 2012-09-14 (Estimated); Status verified 2012-09

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage I prostate cancer; stage IIB prostate cancer; stage IIA prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Gene Expression Profiling; Polymerase Chain Reaction; Reverse Transcriptase Polymerase Chain Reaction; Psychiatric Rehabilitation

INTERVENTIONS:
Behavioral: exercise intervention
Genetic: gene expression analysis
Genetic: polymerase chain reaction
Genetic: proteomic profiling
Genetic: reverse transcriptase-polymerase chain reaction
Other: laboratory biomarker analysis
Other: medical chart review
Other: questionnaire administration
Procedure: psychosocial assessment and care
Procedure: quality-of-life assessment
Procedure: support group therapy
Procedure: therapeutic dietary intervention

SUMMARY:
RATIONALE: Learning about changes in DNA over time in patients with prostate cancer undergoing diet and lifestyle changes may help doctors learn about the long-term effects of these changes on disease progression.

PURPOSE: This clinical trial is studying nutrition and lifestyle changes in patients with previously untreated stage I or stage II prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To measure changes in gene expression in prostate tissue core biopsy samples before and after a low-fat diet and lifestyle intervention in patients with previously untreated stage I or II adenocarcinoma of the prostate.
* To collect health information from these patients to enable better understanding of the long term impact of diet and lifestyle changes on prostate cancer progression.

OUTLINE:

* Intervention phase: Patients are placed on a comprehensive lifestyle change program comprising a low-fat vegan diet, stress management, moderate aerobic exercise, and regular participation in a support group for 3 months.
* Follow-up phase: Patients undergo core tissue biopsies at baseline and at 3 months for genomic and gene expression analysis. Insulin-like growth factor 1 (IGF-1) and selenium-binding protein 1 levels are measured by quantitative reverse transcription-polymerase chain reaction (PCR). Patients also undergo blood sample collection periodically for biomarker analysis, proteomic analysis, and for telomere length and telomerase activity analysis as measured by quantitative PCR and telomerase repeat amplification protocol (TRAP). Blood and urine samples are also collected and stored for future analysis.

Patients complete questionnaires at baseline, at 3 months, and then every 6-12 months for up to 3 years to assess dietary and lifestyle behaviors (exercise, stress management practice, and group support), quality of life, and psychological adjustment. Questionnaires include the Semi-Quantitative Food Frequency Questionnaire; the SF-36 Health Survey; the UCLA Prostate Cancer Index; the Impact of Event Scale; the Memorial Anxiety Scale for Prostate Cancer; the Post Traumatic Growth Inventory; the Mindful Attention Awareness Scale; and the Received Social Support subscale from the Berlin Social Support Scale.

Patients' medical records are reviewed every 6-12 months for up to 3 years to collect information on clinical events and biomarkers (e.g., prostate-specific antigen and Gleason score).

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma (small cell acinar type) of the prostate

  * Has undergone an extended pattern biopsy (defined as 8+ cores) within the past 2 years OR is scheduled to undergo an extended pattern clinical biopsy within 6 weeks of starting study intervention and is willing to undergo 4 additional research core biopsies
  * No more than 33% of biopsy cores positive (> 33% of biopsy cores positive allowed if due to microfoci of adenocarcinoma)
  * No more than 50% of the length of a tumor core involved by carcinoma
* Clinical stage T1 or T2a disease
* Previously untreated disease
* Gleason score ≤ 6 with no pattern 4 or 5 histology (Gleason pattern 4 seen as a microfocus [< 2 mm in length] allowed)
* Prostate-specific antigen (PSA) ≤ 10.0 ng/mL (PSA < 15 ng/mL allowed for patients with benign prostatic hyperplasia or prostatitis)

  * Must have had 3 serum PSA levels performed ≥ 2 weeks apart over the past year to allow calculation of a PSA doubling time

    * No PSA doubling time of < 3 months
* Has chosen watchful waiting as treatment

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy > 3 months
* Living in the greater San Francisco Bay Area
* Willing to make comprehensive lifestyle changes
* Baseline dietary fat intake ≥ 15%
* Able to participate in the exercise portion of this study, as determined by the cardiologist or primary care physician
* No limited exercise tolerance precluding participation in the lifestyle intervention component of this study
* No comprehensive lifestyle change similar to the lifestyle intervention used in this study
* No concurrent uncontrolled illness including, but not limited to, any of the following:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Coronary artery disease requiring a revascularization procedure
  * Cardiac arrhythmia
  * Psychiatric illness/social situation that would limit compliance with study requirements

PRIOR CONCURRENT THERAPY:

* No prior or other concurrent treatment for prostate cancer, including any of the following:

  * Surgery
  * Radiotherapy
  * Hormonal therapy (e.g., leuprolide acetate, bicalutamide, flutamide, goserelin, megestrol acetate, nilutamide, or DES/estrogen)
  * Chemotherapy
  * PC-SPES
  * Investigational agents
* More than 4 weeks since prior and no concurrent finasteride or dutasteride
* More than 4 weeks since prior and no concurrent saw palmetto or any other herbal/nutritional preparation that would affect hormone levels
* More than 4 weeks since prior multivitamin/mineral and/or supplemental soy protein, vitamin E, vitamin C, selenium, fish oil, or any other preparation intended to supplement levels of omega-3 unsaturated fatty acids
* More than 1 month since prior and no concurrent NSAIDs, COX-2-inhibitors, and/or aspirin used for > 7 consecutive days

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2003-09; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Changes in gene expression in prostate tissue core biopsy samples as measured before and after a low-fat diet and lifestyle intervention

SECONDARY OUTCOMES:
Correlation of quality of life changes and adherence to dietary and lifestyle changes with gene expression outcomes
Telomere length and telomerase activity in blood samples in response to the dietary and lifestyle intervention as measured by quantitative polymerase chain reaction and telomerase repeat amplification protocol (TRAP)

CONTACTS AND LOCATIONS:
Overall Officials: Peter R. Carroll, MD, Principal Investigator — University of California, San Francisco

REFERENCES:
- [Result] Ornish D, Lin J, Daubenmier J, Weidner G, Epel E, Kemp C, Magbanua MJ, Marlin R, Yglecias L, Carroll PR, Blackburn EH. Increased telomerase activity and comprehensive lifestyle changes: a pilot study. Lancet Oncol. 2008 Nov;9(11):1048-57. doi: 10.1016/S1470-2045(08)70234-1. Epub 2008 Sep 15. PMID 18799354